CLINICAL TRIAL: NCT04629768
Title: A Study to Evaluate the Effectiveness of Purastat® in the Prevention of Delayed Bleeding After EMR of Non-ampullary Duodenal Lesions
Brief Title: Purastat Prevention Delayed Bleeding Duodenum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. Raf Bisschops (Other)
Collaborators: 3-D Matrix Europe SAS (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Raf Bisschops, Clinical professor, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S63851
Record Dates: First submitted 2020-08-31; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Lesion; Duodenum
Keywords: Purastat; EMR duodenum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duodenal EMR + PuraStat (Other): PuraStat will be applied to the defect after duodenal EMR of the lesion
  Interventions: Device: PuraStat

INTERVENTIONS:
Device: PuraStat — Purastat is applied to the EMR defect

SUMMARY:
PuraStat is a viscous solution of synthetic peptides that provides a physical barrier to facilitate hemostasis. It is indicated for haemostasis in a variety of surgical indications. In this study the efficacy of PuraStat in reducing delayed bleeding following duodenal endoscopic mucosal resection (EMR) will be assessed. PuraStat will be applied to the EMR defect after the resection. The presence of active bleeding or high risk stigma of bleeding will be observed on an esophagogastroduodenoscopy (EGD) performed 1 day after the duodenal EMR. Furthermore the presence of clinical signs of delayed bleeding, other adverse events and the feasibility of PuraStat application will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Duodenal non-ampullary mucosal lesion ≥ 10 mm
* ≥ 18y of age
* Informed consent obtained

Exclusion Criteria:

* Ampulloma
* Submucosal lesion
* Lesion < 10 mm
* >1 lesion resected
* Active use of anticoagulant or antithrombotic medication other than aspirin
* Known clotting disorder
* Inability to give informed consent
* < 18y of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The presence of active bleeding or high risk stigma of bleeding | 1 day after EMR
  On an EGD, performed the day after the duodenal EMR with PuraStat application, the presence of active bleeding or the presence of visible vessels after removal of a blood clot will be observed

SECONDARY OUTCOMES:
The presence of clinical signs of delayed bleeding | 'During hospital stay, assessed up to 10 days' and '30 days after EMR'
  The presence of hematemesis, melena, hemoglobin/hematocrit drop, hypotension or shock will be observed in the patients that had duodenal EMR with PuraStat application.
The presence of other adverse events | 'During hospital stay, assessed up to 10 days' and '30 days after EMR'
  The presence of adverse events like perforation, severe pain, fever… will be observed in the patients that had duodenal EMR with Purastat application
The feasibility of PuraStat application: Amount | During EMR procedure
  The amount of PuraStat will be investigated: Volume in mL
The feasibility of PuraStat application: Ease | During EMR procedure
  The ease of application will be investigated: Questionnaire will be answered by the endoscopist.
The feasibility of Purastat application: Coverage | During EGD procedure
  Is PuraStat covering the resection defect the day after the EMR? This will be investigated by questionnaire that will be answered by the endoscopist who performs the EGD

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Demedts, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium